CLINICAL TRIAL: NCT06014515
Title: Single-tracer Multiparametric PET Imaging
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1921252; 1R01EB033435-01 (NIH)
Record Dates: First submitted 2023-08-07; First posted 2023-08-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects; Cardiovascular Disease
Keywords: total body positron emission tomography
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Participants will undergo two PET/CT scans with two different radiotracers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: PET/CT scans (Experimental): Each subject will undergo a dynamic 18F-FDG PET/CT scan and a dynamic 11C-butanol PET/CT scan on the EXPLORER total-body PET/CT system
  Interventions: Drug: 18F-FDG; Drug: 11C-butanol

INTERVENTIONS:
Drug: 18F-FDG — Each subject will undergo a dynamic 18F-FDG PET/CT scan (this drug is FDA approved) and a dynamic 11C-butanol PET/CT scan (this drug is under an IND) on the EXPLORER total-body PET/CT system. The two scans will be performed on the same day or within a period of up to two weeks depending on subject, imaging agent and scanner availability.
Drug: 11C-butanol — Each subject will undergo a dynamic 18F-FDG PET/CT scan (this drug is FDA approved) and a dynamic 11C-butanol PET/CT scan (this drug is under an IND) on the EXPLORER total-body PET/CT system. The two scans will be performed on the same day or within a period of up to two weeks depending on subject, imaging agent and scanner availability.

SUMMARY:
The overarching goal of this project is to develop and evaluate a single-tracer multiparametric positron emission tomography (PET) imaging solution for simultaneous imaging of blood flow and glucose metabolism using 18F-fluorodeoxyglucose (FDG) alone. The investigators working hypothesis is that quantitative blood flow can be extracted from dynamic 18F-FDG PET data by use of tracer kinetic modeling, in addition to glucose metabolism that 18F-FDG is conventionally used for.

DETAILED DESCRIPTION:
Blood flow and glucose metabolism are two basic but vital physiological processes that are often dysregulated in major diseases. The phenomenon of flow-metabolism mismatch (or coupling) is of broad clinical and research significance. For example, (a) in ischemic cardiomyopathy, which affects several million people in the United States, myocardial flow-metabolism mismatch is clinically used for assessing tissue viability to select patients for surgical revascularization. Decreased blood flow but maintained glucose metabolism suggests the myocytes are still alive (while hibernating) and thus can benefit from revascularization; (b) In oncology, altered blood flow and glucose metabolism are closely related to two hallmarks of cancer - angiogenesis and increased cell metabolism. High metabolism-to-flow ratio may indicate cancer cells are resistant to therapy; (c) In the normal brain, cerebral blood flow and glucose metabolism are often coupled with each other but may become uncoupled in neurodegenerative diseases including Alzheimer's disease. There are critical interests and broad needs for integrated imaging of blood flow and metabolism in both clinical and research applications.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for all research participants:

   * Adults (age ≥ 18 years old)
   * Ability to understand and willingness to sign an informed consent form
   * Ability to adhere to the study visit schedule and other protocol requirements.
   * Willing and able to fast for at least 6 hours before and for the duration of the scan
   * No strenuous exercise for 24 hours prior to being scanned
   * Willing to lie on the scanner bed for up to 60 minutes
   * Free of active COVID-19 symptoms
2. Inclusion Criteria for healthy volunteers only:

   • Free of history of cardiovascular, inflammatory, infections or metabolic diseases that would result in changes in normal tissue perfusion and/or metabolism.
3. Inclusion Criteria for patients with disease:

   * Patients with clinically acute or chronic conditions such as cardiovascular, cardiometabolic, or cardiopulmonary diseases, which may include but are not limited to ischemic heart disease, myocarditis, arrhythmias, heart failure, nonalcoholic fatty liver disease, COVID-related sequala, diabetes, hypertension, or renal disease that would result in changes in normal tissue perfusion and/or metabolism.

Exclusion Criteria:

Participants are not eligible if they meet ANY of the following criteria:

* Self-reported history of dysphoria or anxiety in closed spaces
* Body weight >240 kg due to limitations of the scanner bed
* Pregnant or breast-feeding (due to risks of ionizing radiation; urine pregnancy test will be administered prior to start of each PET/CT session for all participants between 18 to 60 years old who are able to get pregnant, unless documented hysterectomy or bilateral ovarian removal is available)
* Blood glucose greater than 200 as assessed by fingerstick method before injection of 18F-FDG
* Concurrent or prior enrollment in a separate research study involving a PET scan performed within the last 12 months for research purposes only.
* Prisoners
* Any condition that would prevent the understanding or rendering of informed consent.
* Any comorbidity that, in the opinion of the investigator, could compromise protocol objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Blood Flow | during the procedure
  The primary study endpoint is to evaluate if the blood flow estimated with 18F-FDG is quantitatively equal to the blood flow measured with the flow-dedicated tracer 11C-butanol measured in ml/min/g.

SECONDARY OUTCOMES:
Metabolism change when using Butanol | during the procedure
  The secondary endpoint is to assess the changes in metabolism between healthy subjects and patients using Butanol tracer measured in SUV
Metabolism change when using FDG | during the procedure
  The secondary endpoint is to assess the changes in metabolism between healthy subjects and patients using FDG tracer measured in SUV

CONTACTS AND LOCATIONS:
Overall Officials: Guobao Wang, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis EXPLORER Molecular Imaging Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No